CLINICAL TRIAL: NCT06123429
Title: Mindfulness in Hidradenitis Suppurativa
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Arkansas (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 276379
Record Dates: First submitted 2023-10-03; First posted 2023-11-08 (Actual); Last update posted 2024-11-04 (Actual); Status verified 2024-07

CONDITIONS: Hidradenitis Suppurativa
Keywords: Quality of Life; Mindfulness
MeSH Terms: conditions — Hidradenitis Suppurativa | interventions — Mindfulness-Based Stress Reduction

STUDY DESIGN:
Intervention Model Description: Single pilot group, up to 40 patients will enroll and all will receive intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Intervention group (Experimental): All participants enrolled in the study will be enrolled in the Mindfulness-Based Stress reduction course. The MBSR course will consist of weekly sessions lasting two and a half hours, involving lecture, meditation, and self-reflection. The first MBSR course will be ready for 10-12 participants in November 2023. The following course will start every month thereafter. The courses will be held online over Zoom.
  Interventions: Behavioral: Mindfulness Based Stress reduction

INTERVENTIONS:
Behavioral: Mindfulness Based Stress reduction — The MBSR course will consist of weekly sessions lasting two and a half hours, involving lecture, meditation, and self-reflection.
  Mindfulness-Based Stress Reduction (MBSR) is a structured program designed to help individuals manage stress, increase self-awareness, and promote overall well-being. Developed by Dr. Jon Kabat-Zinn in the late 1970s, MBSR combines elements of mindfulness meditation and cognitive-behavioral techniques. MBSR is a comprehensive program that equips individuals with practical skills to better manage stress and enhance their mental and emotional well-being. Its emphasis on mindfulness, self-awareness, and the integration of these practices into daily life makes it a valuable resource for those seeking to reduce stress and improve their overall quality of life.

SUMMARY:
The study will investigate the impact of an 8-week-long Mindfulness-Based Stress Reduction course on quality of life and disease severity in patients with hidradenitis suppurativa (HS).

DETAILED DESCRIPTION:
This is a voluntary 8-week-long, non-medical intervention study for patients with hidradenitis suppurativa (HS). This study will enroll participants in an 8-week-long Mindfulness-Based Stress Reduction course and observed for any changes in validated measures of quality of life. Quality of life scores will be evaluated via multiple surveys including the Dermatology Quality of Life index, HS Quality of Life index, GAD7, and PHQ9. Surveys will be collected Week 1 of 8 week MBSR course intervention; Week 4; End of MBSR Course at week 8; and Week 12. The first goal is to investigate the effectiveness of the addition of mindfulness-based stress reduction (MBSR) intervention to conventional medical treatment on improving mental health in HS participants. The second goal is to assess participant preference for MBSR intervention.

ELIGIBILITY:
Inclusion Criteria:

* This study will only enroll subjects between the ages of 18-years and 89-years of age.
* Diagnosis of HS
* Able to read and comprehend study materials in English, ie: surveys

Exclusion Criteria:

* Those who do not fit inclusion criteria
* Non-English speaking
* Patient who recently began any psychotropic medication within 3 months prior to the baseline evaluation visit.

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2023-10-03 (Actual); Primary Completion 2024-04-30 (Actual); Study Completion 2024-05-30 (Actual)

PRIMARY OUTCOMES:
Dermatology Quality of Life Index (DLQI scores) | Week 1 of 8 week MBSR course intervention; Week 4; End of MBSR Course at week 8; and Week 12
  Change in DLQI scores before and after Mindfulness Based Stress Reduction course.
  DLQI score interpretation:
  0 - 1 no effect at all on patient's life 2 - 5 small effect on patient's life 6 - 10 moderate effect on patient's life 11 - 20 very large effect on patient's life 21 - 30 extremely large effect on patient's life
Generalized Anxiety Disorder (GAD7) | Week 1 of 8 week MBSR course intervention; Week 4; End of MBSR Course at week 8; and Week 12.
  Change in GAD7 scores before and after Mindfulness Based Stress Reduction course. This is calculated by assigning scores of 0, 1, 2, and 3 to the response categories, respectively, of "not at all," "several days," "more than half the days," and "nearly every day." GAD-7 total score for the seven items ranges from 0 to 21. 0-4: minimal anxiety 5-9: mild anxiety 10-14: moderate anxiety 15-21: severe anxiety
Patient Health Questionaire (PHQ9) | Week 1 of 8 week MBSR course intervention; Week 4; End of MBSR Course at week 8; and Week 12.
  Change in PHQ9 scores before and after Mindfulness-Based Stress Reduction course.
  Scoring: add up all checked boxes on PHQ-9 For every 3 Not at all = 0; Several days = 1; More than half the days = 2; Nearly every day = 3 Interpretation of Total Score
  Total Score Depression Severity 1-4 Minimal depression 5-9 Mild depression 10-14 Moderate depression 15-19 Moderately severe depression 20-27 Severe depression

SECONDARY OUTCOMES:
Hidradenitis Suppurativa Quality of Life Index (HiSQOL) | Week 1 of 8 week MBSR course intervention; Week 4; End of MBSR Course at week 8; and Week 12.
  Change in HiSQOL scores before and after Mindfulness-Based Stress Reduction course.
  Grading:
  Not at all = 0 points Slightly = 1 point Moderately = 2 points Very much = 3 points Extremely = 4 points
  0-17 = No effect 18-34 = Small effect 35-51 = Moderate effect 52-68 = Severe effect
  Max score = 68 points

CONTACTS AND LOCATIONS:
Overall Officials: Vivian Shi, MD, Principal Investigator — University of Arkansas
Locations (1):
- UAMS Dermatology Clinic, Little Rock, Arkansas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Vekic DA, Frew J, Cains GD. Hidradenitis suppurativa, a review of pathogenesis, associations and management. Part 1. Australas J Dermatol. 2018 Nov;59(4):267-277. doi: 10.1111/ajd.12770. Epub 2018 Jan 21. PMID 29355905
- [Background] Kouris A, Platsidaki E, Christodoulou C, Efstathiou V, Dessinioti C, Tzanetakou V, Korkoliakou P, Zisimou C, Antoniou C, Kontochristopoulos G. Quality of Life and Psychosocial Implications in Patients with Hidradenitis Suppurativa. Dermatology. 2016;232(6):687-691. doi: 10.1159/000453355. Epub 2017 Jan 5. PMID 28052274
- [Background] Kishimoto S, Watanabe N, Yamamoto Y, Imai T, Aida R, Germer C, Tamagawa-Mineoka R, Shimizu R, Hickman S, Nakayama Y, Etoh T, Sahker E, Carnie MB, Furukawa TA. Efficacy of Integrated Online Mindfulness and Self-compassion Training for Adults With Atopic Dermatitis: A Randomized Clinical Trial. JAMA Dermatol. 2023 Jun 1;159(6):628-636. doi: 10.1001/jamadermatol.2023.0975. PMID 37163257